CLINICAL TRIAL: NCT05269043
Title: SHAPES Advanced Telemonitoring of Patients With COPD in Home Environment
Brief Title: Advanced Telemonitoring of Patients With COPD in Home Environment
Status: Completed | Type: Observational
Sponsor: University Hospital Olomouc (Other)
Responsible Party: Principal Investigator, Ladislav Stanke, Principal Investigator, University Hospital Olomouc
Other Study IDs: SHAPES UC-PT3-COPD
Record Dates: First submitted 2022-01-31; First posted 2022-03-07 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Medimonitor — A digital solution consisting of smartphone/tablet based application gathering data from medical and other devices provided to the patients. These devices are as follows: tablet, smart inhaler, spirometer, blood pressure monitor, pulse oximetry device, particulate matter sensor.

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is one of the leading and rising causes of morbidity and mortality worldwide. The most important etiopathogenetic agent is smoking. However, air-pollution probably also plays a crucial role in the disease development, progression and exacerbations. The multimodal-telemedicine approach may provide a useful tool in the patient follow-up with the aim to reduce disease exacerbation rate and improve the health-related quality of life. The study aims to investigate the effects and utility of advanced telemonitoring in elderly COPD patients. All data will be integrated in a single web-based platform in order to analyse the mutual effects of different conditions and variables.

ELIGIBILITY:
Inclusion Criteria:

* COPD
* ≥ 60 years of age
* Informed written and verbal consent
* Ability to participate in study activities

Exclusion Criteria:

* Active smoking
* Respiratory failure requiring oxygenotherapy or ventilation support
* Severe psychological disturbances
* Absence of collaboration (informed consent)
* Other comorbid pulmonary disease
* Symptomatic heart failure
* Motor neuron diseases (e.g. amyotrophic lateral sclerosis etc.)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic obstructive pulmonary disease.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2022-10-14 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Telemetric spirometry - FVC | 3 month
  Evaluation of telemetric measurement of FVC in home enviroment in COPD patients wih use of mobile spirometer
Telemetric spirometry - PEF | 3 month
  Evaluation of telemetric measurement of PEF in home enviroment in COPD patients wih use of mobile spirometer
Telemetric spirometry - FEV1% | 3 month
  Evaluation of telemetric measurement of FEV1% in home enviroment in COPD patients wih use of mobile spirometer
Telemetric spirometry - FEV1%/FVC ratio | 3 month
  Evaluation of telemetric measurement of FEV1%/FVC ratio in home enviroment in COPD patients wih use of mobile spirometer
Blood oxygen saturation monitoring | 3 month
  Continuous measurement of blood oxygen saturation in the study group.
Particulate matter concentration monitoring | 3 month
  Continuous measurement of both indoor and outdoor air-pollution levels via monitoring of selected parameters (PM1.0, PM2.5, PM4.0, PM10). and some other selected environmental parameters (humidity and temperature) - as well in both outdoor and indoor conditions.
Environmental monitoring | 3 month
  Continuous measurement of selected environmental parameters (humidity and temperature) - in both outdoor and indoor conditions.
Adherence monitoring - rate of inhalations per day | 3 month
  The regular monitoring of the patients' adherence to the inhaled therapy, using FindAir smart inhaler technology. Rate of inhalations per day is measured via special cap mounted on the top of the inhaler which is detecting each activation while pressing the cap. Result is being compared with the amount of inhalations recommended by the physician.
Adherence monitoring - time of inhalation deviation | 3 month
  The regular monitoring of the patients' adherence to the inhaled therapy, using FindAir smart inhaler technology. A specific time of inhalation is being recorded by a special cap mounted on the top of the inhaler which is detecting each activation while pressing the cap. Deviation between recommended time of inhalation and real time of inhalation is being monitored through the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Respiratory Medicine, University Hospital Olomouc, Czech Republic, Olomouc, Czechia

IPD SHARING:
Plan to Share IPD: No